CLINICAL TRIAL: NCT06709781
Title: Cardiovascular Responses in Burn Survivors During Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Craig Crandall, Professor of Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STU_2020-0334_c
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Burn Injury
Keywords: skin graft; thermoregulation; burn survivor; 3rd degree burn injury; human; cooling
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a randomized crossover design study.
  Burn survivors (20% or more burn surface area) and non-burned individuals will perform 60-min of exercise in the heat on two occasions - one being a control (no cooling trial) and one with the implementation of the cooling modality (water spray).
Masking Description: No masking is required as each subject will be exposed to the cooling modality and the control (non-cooling) trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Burned Individuals (Experimental): Non-burned individuals will exercise for 60 minutes in the heat while being exposed to either no cooling or cooling via skin wetting (two trials).
  Interventions: Other: Control (no cooling modalities); Other: Water Spray
- Burn Survivors (20% or more Burn Surface Area burn-injured) (Experimental): Burn survivors with 20% or more BSA (burn surface area) burn-injured will exercise for 60 in the heat while being exposed to either no cooling or cooling via skin wetting (two trials).
  Interventions: Other: Control (no cooling modalities); Other: Water Spray

INTERVENTIONS:
Other: Control (no cooling modalities) — Subjects will exercise for 60 minutes in the heat while being exposed to no cooling modality.
Other: Water Spray — Subjects will exercise for 60 minutes in the heat while being exposed to skin wetting. Skin wetting will be performed by spraying water onto the skin throughout the exercise bout.

SUMMARY:
This project will identify the efficacy of cooling modalities aimed to attenuate excessive elevations in skin and internal body temperatures, and associated indices of cardiovascular stress, during physical activity in well-healed burn survivors. The investigators will conduct a randomized crossover design study. Non-burned control subjects and subjects who experienced burns covering 20% or more of their body surface area will be investigated. Subjects will exercise in heated environmental conditions while receiving no cooling (control) as well as skin wetting.

DETAILED DESCRIPTION:
Within the United States, 500,000+ individuals are enduring the long-term consequences of severe burn injuries covering 20% or more of their body surface area, with upwards to 11,000 individuals experiencing such an injury per year. These burn injuries can severely compromise body temperature regulation, owing to permanent impairments in the primary thermoeffectors necessary to dissipate heat, namely profoundly blunted skin blood flow and sweating responses in the injured skin. The investigators propose that this heat intolerance deters burn survivors from participating in physical activity, including activities of daily living, necessary to avoid the adverse cardiovascular and metabolic sequela of a sedentary lifestyle. Consistent with hypothesis, years after the injury burn survivors have a very low aerobic capacity; greater all-cause mortality rates; greater hospitalization days for circulatory diseases; and suffer from greater incidences of ischemic heart disease, heart failure, diabetes, and cerebrovascular disease (including stroke) relative to matched non-burned cohorts. The primary goal of this project is to identify modalities to attenuate excessive elevations in skin and core body temperatures, and accompanying cardiovascular stress, during physical activity in well-healed burn survivors. The implementation of such modalities will eliminate heat intolerance as a barrier to participation in activities that are necessary to improve/maintain cardiovascular health in this vulnerable population. This project will investigate whether increased skin wetness will restore otherwise impaired evaporative cooling of well-healed burn survivors, with the extent of that improvement predicated on the environmental conditions and the percentage of body surface area burned.

ELIGIBILITY:
Inclusion Criteria: Non-Burned Individuals

* Healthy male and female subjects
* 18-65 years of age.
* Free of any underlying medical conditions

Exclusion Criteria: Non-Burned Individuals

* Any burn-related injuries resulting in at least one night of hospitalization.
* Heart disease or any other chronic medical condition requiring regular medical therapy including cancer, diabetes, and hypertension.
* Abnormalities detected on routine screening
* Individuals who participate in a structured aerobic exercise training program at moderate to high intensities.
* Current smokers, as well as individuals who regularly smoked within the past 3 years.
* Body mass index of greater than 30 kg/m^2.
* Pregnant individuals

Inclusion Criteria: Burn Survivors

* Healthy male and female subjects
* 18-65 years of age.
* Free of any underlying medical conditions
* Having a burn injury covering 20% or more of the participant's body surface area; at least 50% of those burn injuries must be full thickness that required skin grafting.
* Participants must have been hospitalized due to the burn injury for a minimum of 15 days

Exclusion Criteria: Burn Survivors

* Any burn-related injuries resulting in at least one night of hospitalization.
* Heart disease or any other chronic medical condition requiring regular medical therapy including cancer, diabetes, and hypertension.
* Abnormalities detected on routine screening
* Individuals who participate in a structured aerobic exercise training program at moderate to high intensities.
* Current smokers, as well as individuals who regularly smoked within the past 3 years.
* Body mass index of greater than 30 kg/m^2.
* Pregnant individuals
* Extensive unhealed injured skin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Core Temperature (°C) During Control Intervention | At 0 minutes and 60 minutes into the intervention.
  The subject's core body temperature will be measured from gastrointestinal or rectal temperature measures.
Change in Core Temperature (°C) During Water-Spray Intervention | At 0 minutes and 60 minutes into the intervention.
  The subject's core body temperature will be measured from gastrointestinal or rectal temperature measures.

SECONDARY OUTCOMES:
Skin Temperature (°C) Following Control Intervention | At 60 minutes into the intervention.
  The subject's skin temperature will be measured from small temperature sensitive electrodes attached to the participant's skin.
Skin Temperature (°C) Following Water-Spray Intervention | At 60 minutes into the intervention.
  The subject's skin temperature will be measured from small temperature sensitive electrodes attached to the participant's skin.
Heart Rate Following Control Intervention | At 60 minutes into the intervention.
  The subject's heart rate will be measured from ECG electrodes attached to the participant.
Heart Rate Following Water-Spray Intervention | At 60 minutes into the intervention.
  The subject's heart rate will be measured from ECG electrodes attached to the participant.
Mean Arterial Blood Pressure Following Control Intervention | At 60 minutes into the intervention.
  The subject's mean arterial blood pressure will be measured using a standard arm blood pressure cuff.
  Mean Arterial Pressure (MAP) is a common physiological measure calculated by adding the diastolic blood pressure value to one third of the difference between the systolic (SBP) and diastolic (DBP) blood pressure values.
  MAP = DBP + 1/3(SBP - DBP)
Mean Arterial Blood Pressure Following Water-Spray Intervention | At 60 minutes into the intervention.
  The subject's mean arterial blood pressure will be measured using a standard arm blood pressure cuff.
  Mean Arterial Pressure (MAP) is a common physiological measure calculated by adding the diastolic blood pressure value to one third of the difference between the systolic (SBP) and diastolic (DBP) blood pressure values.
  MAP = DBP + 1/3(SBP - DBP)

CONTACTS AND LOCATIONS:
Overall Officials: Craig G Crandall, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Institute for Exercise and Environmental Medicine - Texas Health Presbyterian Hospital Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No